CLINICAL TRIAL: NCT03141164
Title: Peripheral Vision Training Study
Acronym: PVTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kristina M Visscher, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: X101022014
Record Dates: First submitted 2017-04-28; First posted 2017-05-04 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Visual Impairment; Cognitive Change
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Masking Description: Computerized training for all groups. This is a pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): Computerized vision training
  Interventions: Other: computerized training
- Control (Sham Comparator): Sham
  Interventions: Other: computerized training

INTERVENTIONS:
Other: computerized training — Computerized training

SUMMARY:
This study will train participants (young people and older adults) to do a visual task, and will assess whether this results in changes in behavioral assessments. In some participants, we will be also testing whether MRI measures (cortical thickness, functional connectivity) change with training.

ELIGIBILITY:
Inclusion criteria:

* Right handed individuals
* Aged 19-89
* In good health as self-reported or visual impairments due to partial vision loss
* Normal or corrected-to-normal vision with contact lenses or visual impairments due to partial vision loss

Exclusion criteria:

* Younger than 18 or older than 89
* Being hearing-impaired
* Not in good health except due to partial vision loss
* Having a previous serious head injury or neurological disorder, or loss of consciousness for more than 2 minutes
* Having hallucinations or delusions
* Having a current or past history of a substance abuse disorder
* Currently taking psychoactive medications

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
scores on acuity tests | baseline
  scores on acuity tests
scores on acuity tests | immediately following training
  scores on acuity tests
scores on spatial attention tests | baseline
  scores on spatial attention tests
scores on spatial attention tests | immediately following training
  scores on spatial attention tests

SECONDARY OUTCOMES:
Changes in cortical thickness | baseline and immediately following training
  Increases in cortical thickness in areas corresponding to trained visual field
Changes in functional connectivity | baseline and immediately following training
  Changes in functional connectivity of areas corresponding to trained visual field

CONTACTS AND LOCATIONS:
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No